CLINICAL TRIAL: NCT04240522
Title: Prospective Longitudinal Observational Research Study to Investigate the Remission of Atopic Dermatitis and Associated Allergic Diseases
Brief Title: Prospective Longitudinal Observational Research in Atopic Dermatitis
Acronym: ProRaD
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: ProRaD
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis; Asthma; Atopic Dermatitis and Related Conditions
Keywords: Eczema; Dermatitis; Atopy
MeSH Terms: conditions — Dermatitis, Atopic; Asthma; Eczema; Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples, Microbiom swabs Ski biopsy (selcted cases)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atopic dermatitis (AD) is a frequent chronic relapsing inflammatory skin disorder, characterized by intensely itchy eczema. AD usually starts within the first 2 years of life. In 30 - 60% of children, inflammation spreads onto other body surfaces such as the gastrointestinal tract, the respiratory tract, and the conjunctives within a few years. This sequence is called atopic march.

Atopic dermatitis and associated atopic diseases are more frequent in families, suggesting a genetic predisposition. However, the underlying factors such as genetic phenotype, environmental factors, or life style which cause or worsen an existing allergic disease are not understood yet. Affected people suffer from recurrent flares that result in significantly impaired quality.

This study will collect clinical and laboratory data to elucidate immunotolerance and preventiv stategies with the aim to develop new and individual treatment options of atopic diseases.

DETAILED DESCRIPTION:
Primary Objetive:

In the planned project, the main objective is to identify endogenous (e.g. immunological and molecular factors) and exogenous factors (e.g. environmental, socioeconomic and microbial factors) that influence the course and remission of AD. More specifically to identify factors that are significantly different between patients that have or do not have remission from AD.

Secondary Objective:

(i) To identify endogenous and exogenous factors such as immunological, molecular and microbial factors to separate subgroups of patients (endotypes) with distinct local and systemic inflammatory responses.

(ii) To identify potential biomarkers predicting the individual clinical course of AD and other atopic diseases including asthma, food allergy and allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 - 85 years
* Diagnosis of AD and/or another disease of the atopic group (i.e. allergic rhinitis, allergic asthma, food allergy)
* The inclusion of patients in this study is independent from the current therapy. During the study all patients will be kept on a therapy that is medically indicated

The inclusion criteria for healthy controls in this study are as follows:

* Age 0 - 85 years
* No diagnosis or history of allergic disease
* The inclusion of patients in this study is independent from the current therapy. During the study all patients will be kept on a therapy that is medically indicated

Written consent will be obtained after detailed information of the study was given to the participant.

Exclusion Criteria

- Unable to give consent or refusal to participate in the study

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with atopic dermatits, any other allergic diseases and /or healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2031-03-30 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
Remission of atopic dermatitis and associated allergic diseases | 5 years
  Prospective observational study

SECONDARY OUTCOMES:
Endogenous and exgogenouse factors that influence and predict the course of AD. | 5 years
  Prospective observational study
Identification of potential biomarkers predicting the course of AD | 5 years
  Prospective observational study

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy Unit, Dept. of Dermatology, Unviersity Hosptial of Zurich, Zurich, Canton of Zurich, Switzerland